CLINICAL TRIAL: NCT01415206
Title: Extended Care Treatment of Multiple Risk Behaviors in Complex Patients
Brief Title: The Total Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-01298; P50DA009253 (NIH)
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Risk Reduction Behavior
Keywords: Behavioral changes; Multiple risks
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended Staging Health Risk Intervention (S-HRI) (Experimental): The S-HRI provides feedback on participants' stages of change for each risk and the single most important step they can take to begin progressing. A counselor will review the report with participants and provide motivational interviewing (MI) coaching and referrals to relevant behavior change services. Repeated computer and individual counseling contacts at baseline, 3, 6 and 12 months follow-up are designed to support participants through the process of changing multiple risk behaviors.
  Interventions: Behavioral: Extended Staging Health Risk Intervention (S-HRI)
- Usual Care (Other): Participants in the usual care condition will complete the core assessments and the Staging Health Risk Assessment (S-HRA) online at baseline, 3, 6, 12, and 18 months follow-up but will not meet with the study MI coach and will NOT receive any feedback or printed report until the 18-month follow-up.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Extended Staging Health Risk Intervention (S-HRI) — The S-HRI provides feedback on participants' stages of change for each risk and the single most important step they can take to begin progressing. A counselor will review the report with participants and provide motivational interviewing (MI) coaching and referrals to relevant behavior change services. Repeated computer and individual counseling contacts at baseline, 3, 6 and 12 months follow-up are designed to support participants through the process of changing multiple risk behaviors.
  Arms: Extended Staging Health Risk Intervention (S-HRI)
Behavioral: Usual Care — Participants in the usual care condition will complete the core assessments and the S-HRA online at baseline, 3, 6, 12,and 18 months follow-up but will not meet with the study MI coach and will NOT receive any feedback or printed report until the 18-month follow-up.
  Arms: Usual Care

SUMMARY:
This study is a randomized, controlled, multiple risk intervention pilot study evaluated with clients recruited from VA Medical Center Substance Abuse Programs. The intervention combines an innovative online system with interpersonal MI-based coaching delivered in 4 sessions over 12-months time.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are: at least 18 years of age, enrolled in the San Francisco Veteran Affairs Medical Center (SF VAMC) Substance Abuse Programs, residing in the San Francisco Bay Area and not planning to relocate out of the area in the next 18 months. For patients in the Day Hospital, we will wait until they have completed one week of treatment before approaching for study involvement, as the first week is the most intensive for services.

Exclusion Criteria:

* Exclusion criteria are: unstable psychiatric disorder and severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06-02 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Client engagement with behavior change service referrals | Up to18 months follow-up.

SECONDARY OUTCOMES:
Behavioral changes in multiple risks | up to 18 months follow-up.
Improvements in health-related quality of life at 3, 6, 12, and 18 months follow-up. | up to 18 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Judith J Prochaska, PhD, MPH, Principal Investigator — Stanford University
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States